CLINICAL TRIAL: NCT06140472
Title: Effectiveness of the PHOENIX Smartphone Application on the Nursing Management of Craving in Patients With Addictive Disorders Followed on an Outpatient Basis
Brief Title: PHOENIX: Craving Management Smartphone Application
Acronym: PHOENIX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier St Anne (Other)
Collaborators: Direction Générale de l'Offre de Soins (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: D19-P019
Record Dates: First submitted 2019-09-27; First posted 2023-11-20 (Actual); Last update posted 2023-11-20 (Actual); Status verified 2023-11

CONDITIONS: Craving
Keywords: Addiction; Craving; Mobile application; Craving management
MeSH Terms: conditions — Behavior, Addictive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phoenix application (Active Comparator): Specific individualized nurse follow-up using the PHOENIX application.
  Interventions: Behavioral: Phoenix
- Journal de bord (Sham Comparator): Regular nursing follow-up, with the use of an electronic journal.
  Interventions: Behavioral: Journal de bord

INTERVENTIONS:
Behavioral: Phoenix — Specific individualized nurse follow-up using the PHOENIX application.
  Arms: Phoenix application
Behavioral: Journal de bord — Regular nursing follow-up, with the use of an electronic journal.
  Arms: Journal de bord

SUMMARY:
The objective of this study is to evaluate the effectiveness of the addition of nursing follow-up and the PHOENIX application, a personalized and self-adaptive Smartphone application, on the management of craving in patients with addictive disorders followed on an outpatient basis.

DETAILED DESCRIPTION:
Addictive disorders are a public health priority. The management of addictive disorders aims to reduce addictive behaviour or abstinence, implying that the patient can overcome the urge to engage in this behaviour, a symptom called craving.

Craving, as a major motivational substrate for addictive behaviour, is a preferred therapeutic target for the management of addictive disorders. However, to date, there are no fully effective drugs or psychological interventions. Smartphone applications seem to have an interest in this context, with many advantages: accessibility, anonymity, ease of access and low cost. Sainte Anne's Hospital Moreau de Tour facility (Paris, France) was one of the pioneering centres in the management of addictive disorders. The nursing team has developed expertise in this field. Patients report difficulties to nurses about managing their craving on their own, and ask for more frequent interviews or even daily support. During practice analysis meetings, caregivers sought innovative solutions to optimize this care. Our team has designed the PHOENIX application, which allows us to support patients in real time who wish to reduce or stop their addictive behaviours. Used between two consultations, it targets craving, without being specific to a product or addictive behaviour. When the patient has a craving, PHOENIX identifies the situation and proposes the most appropriate strategy to avoid using. Strategies are personalized and self-adaptive. The application allows caregivers to monitor patients' progress and progress.

Hypothesis of this study: The PHOENIX application used as a complement to nursing care will allow a better management of craving and a decrease in relapses compared to usual care (usual care: multidisciplinary care including nursing care).

ELIGIBILITY:
Inclusion Criteria:

* Being 18 and 65 years old, any sex
* Speak and read French
* Have a Smartphone (Android operating system or IOS)
* Present an evaluated addictive disorder in a structured clinical interview (MINI, adapted to the criteria of DSM-5: substance use disorder according to DSM-5 and bulimia nervosa; National Opinion DSM Screen (NODS), adapted to the criteria of DSM-5: pathological gambling; NODS, adapted to the diagnostic criteria proposed by Carnes: sexual addiction ; MINI)
* Be followed on an outpatient basis
* Prior informed written consent of the patient or his or her legal representative
* Benefit from a French social protection system

Exclusion Criteria:

* Have a current untreated and/or unstabilized psychiatric disorder (assessed by MINI)
* Have a severe cognitive impairment assessed during the clinical interview, which does not allow you to focus your attention or use the working memory required by the application.
* Pregnant or breastfeeding women
* Participant in another clinical trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2019-12-11 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
median craving intensity at 6 months | 6 months visit
  Measurement of craving intensity with an analog visual scale (AVS) between 0 (no craving) and 10 (maximum imaginable craving), informed during craving episodes by the patient via the PHOENIX application or the electronic journal. Over the last 30 days before the visit at 6 months

SECONDARY OUTCOMES:
Number of cravings | 0,3,6 and 12 months visit
  The cravings will be informed by the patient during craving episodes via the PHOENIX application or the electronic journal
Daily frequency of cravings | 0,3,6 and 12 months
  The cravings will be informed by the patient during craving episodes via the PHOENIX application or the electronic journal
Median of the intensity of the cravings | 0, 3, and 12 months visit
  Measurement of craving intensity with an analog visual scale (AVS) between 0 (no craving) and 10 (maximum imaginable craving), informed during craving episodes by the patient via the PHOENIX application or the electronic journal. Over the last 15 days before the visit at 0, 3 and 12 months
Number of addictive behavioural episodes | 0,3,6 and 12 months
  Addictive behaviors will be informed via the phoenix application or the electronic journal
Frequency of addictive behavioural episodes | 0,3,6 and 12 months
  Addictive behaviors will be informed via the phoenix application or the electronic journal
Type of addictive behavioural episodes | 0,3,6 and 12 months visit
  Addictive behaviors will be informed via the phoenix application or the electronic journal
Severity of addictive disorder: addictive substance disorder or pathological gambling | 0,3,6 and 12 months
  Severity of the disorder assessed by the number of diagnostic criteria for addictive substance disorder or pathological gambling on the Diagnostic and Statistical Manuel of mental disorders (DSM-5).
Severity of addictive disorder: Yale Food Addiction Scale (YFAS) food addiction score for bulimia nervosa | 0 and 12 months visit
  Severity of the food addiction for bulimia nervosa is assessed by the Yale Food Addiction Scale (YFAS).
  The YFAS assesses addiction-like eating of palatable foods based on the 11 diagnostic criteria for substance use disorder in the Diagnostic and Statistical Manual of Mental Disorders (DSM-5). No Food Addiction = 0-1 symptoms/score; Mild Food Addiction = 2 or 3 symptom/score; Moderate Food Addiction = 4 or 5 symptom/score; Severe Food Addiction = 6 or higher symptom/score
Severity of addictive disorder: sexual addiction (Carnes criteria) | 0,3,6 and 12 months visit
  Severity of the disorder assessed by the number of positive responses in the Carnes criteria. Carnes criteria consists of 25 yes/no questions. If the answer is "yes" to 13 or more questions, the patient can be diagnosed as a sex addict (range: 0-25).
Impulsivity (UPPS scale) | 0,3,6 and 12 months
  Impulsivity is assessed using the UPPS scale (Urgency, Premeditation (lack of), Perseverance (lack of), Sensation seeking. The UPPS impulsivity scale is a 45-item self-questionnaire that measures impulsivity by exploring: urgency (12 items: range 12-48), lack of forethought (11 items; range:11-44), lack of perseverance (10 items; range:10-40) and sensation seeking (12 items; range:12-48). For each subdimension, a high score indicates a high level of impulsivity.
Number of strategies to deal with craving according to the type of addictive behaviour | 0,3,6 and 12 months
  The strategies will be provided through the application or the electronic journal
Multidimensional evaluation of coping (Brief Cope scale by Muller and Spitz) | 0,3,6 and 12 months
  The multidimensional evaluation of coping is carried out using the Brief Coping Orientation to Problems Experienced (Brief COPE) ,28-item self-questionnaire. The Brief COPE contains 28 statements and 14 scales, each consisting of 2 statements. It is a self-administered questionnaire. It is available in 2 formats: 1) dispositional, which is designed to assess how people habitually respond to stressful situations, and 2) situational, which is designed to assess how people responded to a specific event or context that has recently become a source of stress. Only the verb tense varies between statements in the two formats.
  The respondent uses a 4-point scale to give his/her answer to each statement: 1 - not at all; 2 - a little; 3 - a lot; 4 - completely.
  The answers obtained are added together for each scale. Higher scores on a scale indicate greater use of this coping mechanism.
Anxiety: Beck's inventory for anxiety (BAI) | 0,3,6 and 12 months
  The anxiety assessment is carried out using Beck's inventory for anxiety (BAI). The Beck Anxiety Inventory (BAI) is a 21-question multiple-choice self-report inventory used to measure the severity of anxiety. The questions used in this measure ask to describe common symptoms of anxiety that the subject has experienced in the last week (including the day on which the measure is taken).
  The BAI contains 21 questions, each answer being scored on a scale value of 0 (not at all) to 3 (severely). Higher total scores indicate more severe anxiety symptoms.
  The standardized cutoffs are:
  0-7: Minimal 8-15: Mild 16-25: Moderate 26-63: Severe
Depression: Beck's depression inventory | 0,3,6 and 12 months
  The Beck Depression Inventory (BDI), is a multiple-choice self-report inventory for measuring the severity of depression.
  The BDI, consisted of twenty-one questions about how the subject has been feeling in the last week. Each question had a set of at least four possible responses, ranging in intensity:
  (0) I do not feel sad
  1. I feel sad.
  2. I am sad all the time, and I cannot snap out of it.
  3. I am so sad or unhappy that I cannot stand it.
  When the test is scored, a value of 0 to 3 is assigned for each answer, and then the total score determines the depression's severity. The standard cut-off scores were as follows:
  0-9: indicates minimal depression 10-18: indicates mild depression 19-29: indicates moderate depression 30-63: indicates severe depression. Higher total scores indicate more severe depressive symptoms.
Quality of life: World Health Organization Quality of Life (WHOQOL 26 scale) | 0,3,6 and 12 months
  The World Health Organization Quality of Life (WHOQOL26) assesses subjective health-related quality of life in a 26-item self-administered questionnaire.
  The WHOQOL26 scale investigates the quality of life in four domains: physical health (7 items), psychological health (6 items), social relationships (3 items) and environmental health (8 items); it also contains QOL and general health items. Each item of the WHOQOL26 is scored on a five-point ordinal scale. The scores are then linearly transformed into a 0-100 scale.
Self-esteem (Coopersmith inventory) | 0,3,6 and 12 months
  The Coopersmith's Self-Esteem Inventory assesses general, professional, social and family self-esteem; the total is the sum of these four components. The test comprises 58 items; the responses are "looks like me" or "doesn't look like me." The score is composed of several subscales: General (26 items), Social (8 items), Professional (8 items), Family (8 items) and Lie (8 items). The total score (50 items) is obtained by summing the General, Social, Professional and Family subscales. The Lying scale is more of a social desirability scale used to assess patient authenticity in general assessment.
Use of healthcare related to addictive disorder: Hospitalisation | 0,3,6 and 12 months
  Number of hospitalization days related to addiction
Use of healthcare related to addictive disorder: emergency department accesses | 0,3,6 and 12 months
  Number of emergency department accesses related to addiction

CONTACTS AND LOCATIONS:
Overall Officials: Chloe Lucet, PH, Principal Investigator — Centre Hospitalier St Anne
Locations (2):
- France (2):
  - Hospices Civiles de Lyon, Lyon
  - CHU de Nantes, Nantes